CLINICAL TRIAL: NCT06400485
Title: First-in-Human, Phase 1 Study of AMT-676 in Patients With Advanced Solid Tumors
Brief Title: AMT-676 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Multitude Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT-676-01
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMT-676 Dose escalation (Experimental): Drug- AMT-676 Dosage level: AMT-676 will be administered as an intravenous (IV) infusion. Dosage form: Vial Route of administration: Intravenous Infusion
  Interventions: Drug: AMT-676

INTERVENTIONS:
Drug: AMT-676 — Participants will receive AMT-676 administered intravenously. Participants will be observed for first instance of dose limiting toxicities (DLT).

SUMMARY:
This is a first-in-human, non-randomized, open-label, multicenter Phase 1 study will evaluate the Maximum tolerated dose (MTD)/the recommended Phase 2 Dose (RP2D), safety, tolerability, anti-drug activity, pharmacokinetics, pharmacodynamics and immunogenicity of AMT-676 in Patients with Advanced Solid Tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients must be willing and able to sign the ICF, and to adhere to the study visit Schedule and other protocol requirements.
2. Age ≥18 years (at the time consent is obtained).
3. Patients with pathologically confirmed unresectable advanced solid tumor. Preferred tumor types include colorectal cancer, gastric cancer, esophageal adenocarcinoma, cholangiocarcinoma, pancreatic ductal cancers, and neuroendocrine tumors.
4. Patients who have undergone at least one systemic therapy and have radiologically or clinically determined progressive disease during or after most recent line of therapy, and for whom no further standard therapy is available, or who are intolerable to standard therapy.
5. Patients must have at least one measurable lesion as per RECIST version 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. Life expectancy ≥3 months.
8. Patients must have adequate organ function
9. Women of child-bearing potential (WCBP) must have a negative serum pregnancy test.
10. Male patients must agree to use a latex condom, even if they had a successful vasectomy, while on study treatment and for at least 6months after the last dose of the IMP.
11. Male patients must agree not to donate sperm, and female patients must agree not to donate eggs, while on study treatment and for at least 3 months and 6 months, respectively after the last dose of the IMP.
12. Availability of tumour tissue sample (either an archival specimen or a fresh biopsy material) at screening.

Key Exclusion Criteria:

1. Prior treatment with any agent for the same target or ADC based on topoisomerase I inhibitor.
2. Central nervous system (CNS) metastasis
3. History of Steven's Johnson's syndrome or toxic epidermal necrolysis syndrome.
4. Persistent toxicities from previous systemic anti-neoplastic treatments of Grade >1.
5. Systemic anti-neoplastic therapy within five half-lives or21 days, whichever is shorter, prior to first dose of the IMP.
6. Radiotherapy to lung field at a total radiation dose of ≥20 Gy within 6 months, wide-field radiotherapy (e.g., >30% of marrow-bearing bones) within 28 days.
7. Major surgery (not including placement of vascular access device or tumor biopsies) within 28 days prior to first dose of the IMP, or no recovery from side effects of such intervention.
8. Significant cardiac disease, such as recent (within months prior to first dose of the IMP) myocardial infarction or acute coronary syndromes (including unstable angina pectoris), congestive heart failure (New York Heart Association class III or IV), uncontrolled hypertension (SBP ≥ 160mmHg or DBP ≥ 100mmHg), uncontrolled cardiac arrhythmias.
9. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or current ILD/pneumonitis, or suspected ILD/pneumonitis (e.g., idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, etc.) or other lung disease significantly impacting lung function at baseline.
10. History of thromboembolic or cerebrovascular events, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis, or pulmonary emboli within six months prior to first dose of the IMP.
11. Acute and/or clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV)
12. Administration of a live vaccine within 28 days prior to the administration of the first dose of the IMP.
13. Patients requiring concurrent treatment of strong inhibitors or inducers of cytochrome P450 3A4 or 1A2 enzyme (CYP3A or CYP1A2) within 2 weeks prior to the first dose and during the study treatment.
14. Known or suspected severe allergy/hypersensitivity (resulting in treatment discontinuation) to monoclonal antibodies.
15. Known or suspected intolerance to the components of the IMP.
16. Concurrent participation in another investigational therapeutic clinical trial.
17. Patients with known active alcohol or drug abuse.
18. Pregnant or breast-feeding females
19. Mental or medical conditions that prevent the patient from giving informed consent or complying with the trial or other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with the study participation or the IMP administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrolment in this study.
20. Prior history of malignancy other than inclusion diagnosis within five years prior to first dose of the IMP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | 30 days after the last dose of IMP
  The RP2D will be determined using dose limiting toxicities (DLTs) and all other available study data
Maximum Tolerated Dose (MTD) | 30 days after the last dose of IMP
  The MTD will be determined using DLTs
Type, incidence and severity of Adverse Events | 30 days after the last dose of IMP
  Safety and tolerability profile assessed by the Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Maximum observed concentration (C[max]) | 30 days after the last dose of IMP
  Pharmacokinetic profile characterized by the maximum observed concentration (C[max]) of AMT-676
Time to maximum concentration (Tmax) | 30 days after the last dose of IMP
  Pharmacokinetic profile characterized by the time to maximum concentration (Tmax) of AMT-676
Area under the curve (AUC) | 30 days after the last dose of IMP
  Pharmacokinetic profile characterized by the area under the curve (AUC) of AMT-676
Terminal half-life (t[1/2]) | 30 days after the last dose of IMP
  Pharmacokinetic profile characterized by the terminal half-life (t[1/2]) of AMT-676
Concentration of anti-drug antibodies (ADA) | 30 days after the last dose of IMP
  Immunogenicity profile characterized by concentration of ADAs
Overall Response Rate (ORR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | 30 days after the last dose of IMP
  Proportion of patients achieving Complete Response (CR) or Partial Response (PR)
Disease Control Rate (DCR) according to the RECIST v1.1 | 30 days after the last dose of IMP
  Proportion of patients achieving CR, PR or Stable Disease (SD)
Progression-free Survival (PFS) | 30 days after the last dose of IMP
  Time from date of start of treatment to date of the first progression or death, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (13):
- American Samoa (3):
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - John Hopkins Sidney Kimmel Comprehensive Cancer Center, Philadelphia, Pennsylvania
  - South Texas Accelerated Research Therapeutics (start) San Antonio, San Antonio, Texas
- Australia (5):
  - SCIENTIA Clinical Research Ltd, Randwick, New South Wales
  - Macquarie University Hospital, Macquarie, New South wWales
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Cabrini Hospital, Melbourne, Victoria
  - Linear Research, Nedlands, Western Australia
- China (5):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No